CLINICAL TRIAL: NCT00359411
Title: Genetic Studies of the X-Linked Lymphoproliferative Disease
Brief Title: Genetic Studies of X-linked Lymphoproliferative Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960085; 96-I-0085
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-01

CONDITIONS: X-Linked Lymphoproliferative Disease; Lymphoproliferative Disease; Genetic Diseases, X-Linked
Keywords: Epstein-Barr Virus; B-Cell Lymphoma; Herpes Virus; Infectious Mononucleosis
MeSH Terms: conditions — Lymphoproliferative Disorders; Genetic Diseases, X-Linked; Epstein-Barr Virus Infections; Lymphoma, B-Cell; Infectious Mononucleosis

SUMMARY:
This study will study the effects of the gene on the X chromosome that is associated with X-linked lymphoproliferative disease (XLPD)-an inherited disease affecting the immune system-on the function of the immune system. XLPD has been linked to an abnormality in a specific region of the X chromosome (one of 23 chromosome pairs that contain the genes that determine a person's hereditary makeup). The disease may develop after infection with the Epstein-Barr virus (EBV). EBV affects more than 95 percent of people in the United States. It usually does not cause any symptoms in children. In adolescents and adults, however, EBV can cause infectious mononucleosis and sometimes lymphoproliferative disease, such as XLPD. In these diseases lymph tissues, such as lymph nodes, may become enlarged and immune function (infection-fighting ability) impaired. This study will compare DNA from patients with XLPD with that of their unaffected relatives, of patients with other lymphoproliferative diseases and of normal controls.

Patients of any age with XLPD, their unaffected relatives 18 years of age and older, and patients with other lymphoproliferative diseases may participate in this study.

Blood samples will be collected from all participants to study the effects of the gene on the X chromosome that appears to be abnormal in XLPD on the function of the immune system. In a 6-week period, no more than 100 milliliters (about 7 tablespoons) of blood will be drawn from adults and no more than 1 ml (1/6 teaspoon) of blood per pound of body weight from children. Blood from patients with XLPD and their relatives will also be tested for HLA type (similar to blood type testing) and the ability of HLA-matched cells from patients and relatives to interact will be examined.

...

DETAILED DESCRIPTION:
Males with the X-linked ymphoproliferative disease (XLPD) have a marked susceptibility to Epstein-Barr virus (EBV) disease. These boys develop very severe disease associated with infectious mononucleosis; others develop hypogammaglobulinemia or B cell lymphomas. Recent studies have linked the disease to a region of the X-chromosome. The purpose of this study is to determine the function of the gene responsible for XLPD. Blood samples or discarded tissues (e.g. previous biopsy or autopsy material) from patients with XLPD and their relatives will be analyzed to determine the precise genetic defect associated with the disease. Blood samples or discarded tissues from other patients with EBV-associated lymphoproliferative diseases and blood samples from normal individuals will be obtained to serve as controls. Knowledge gained from this study should provide important insights into the immunologic control of EBV lymphoproliferative disease associated with congenital or acquired immunodeficiency. In addition, identification of the molecular mechanisms for these diseases may provide clues to other EBV-associated diseases including nasopharyngeal carcinoma, Burkitt lymphoma, and Hodgkin's disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients known to have XLPD and their relatives will be recruited from families who have enrolled in a national XLPD registry.

All racial and ethnic groups will be considered.

To be considered having XLPD, a patient must be a male who has had:

* severe infectious mononucleosis, or
* acquired hypogammaglobulinemia following infectious mononucleosis, or
* nonHodgkin's lymphoma, or
* hyper-IgM or an IgG subclass deficiency with evidence of linkage to the DXS42 locus

and

have no other known immunocompromising condition and belong to a family in which another related male has had one or more of the above listed phenotypes.

EXCLUSION CRITERIA:

Known HIV infection in any patient with XLPD or their relative (blood will not be tested for HIV), complicating medical or psychiatric conditions in unrelated controls.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1996-05-22; Study Completion 2010-02-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Purtilo DT, Cassel CK, Yang JP, Harper R. X-linked recessive progressive combined variable immunodeficiency (Duncan's disease). Lancet. 1975 Apr 26;1(7913):935-40. doi: 10.1016/s0140-6736(75)92004-8. PMID 48119
- [Background] Skare JC, Milunsky A, Byron KS, Sullivan JL. Mapping the X-linked lymphoproliferative syndrome. Proc Natl Acad Sci U S A. 1987 Apr;84(7):2015-8. doi: 10.1073/pnas.84.7.2015. PMID 2882515
- [Background] Cohen JI. Epstein-Barr virus lymphoproliferative disease associated with acquired immunodeficiency. Medicine (Baltimore). 1991 Mar;70(2):137-60. doi: 10.1097/00005792-199103000-00005. PMID 1848644